CLINICAL TRIAL: NCT03796065
Title: Addressing Mental Health Disparities in Refugee Children Through Family and Community-based Prevention: A CBPR Collaboration and Hybrid Implementation Effectiveness Trial
Brief Title: Addressing Mental Health Disparities in Refugee Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18.251.01
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Family Research
Keywords: refugees; parental self-efficacy; family communication; family connectedness; refugee youth; youth functioning; integration

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a Randomized Controlled Trial among Somali Bantu and Bhutanese families (N=300; 150 per group). Half of the families will be randomized to receive the FSI-R and half will be randomized to the control condition where the participants will receive Treatment as Usual (TAU).
Who Masked: Care Provider
Masking Description: The Research Assistants (RAs) who will collect both qualitative and quantitative data will be blind to the condition in which study participants are randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FSI-R Treatment (Experimental): Families randomized into the FSI-R Treatment arm will receive the 10-module Family Strengthening Intervention in addition to any outside services or programs they are participating in.
  Interventions: Behavioral: FSI-R Treatment
- FSI-R Control (No Intervention): Families randomized into the FSI-R Control arm will not receive the FSI-R treatment. Instead, they will continue with their usual care, referred to as Treatment as Usual (TAU).

INTERVENTIONS:
Behavioral: FSI-R Treatment — The FSI-R involves a series of separate and joint meetings with parents and children to discuss challenges the family has faced and the strengths that helped them make it through past challenging times. Additional psychoeducation on mental health and promoting resilience along with coaching to enhance parenting skills is provided throughout and may be tailored to family needs. The FSI-R provides a shared space for refugee families both to recognize their strengths and to problem-solve in a more collective way on family challenges and shared hopes for the future. The FSI-R is delivered in the home, by a trained interventionist, over the course of 10-modules.
  Other Names: Family Strengthening Intervention for Refugees
  Arms: FSI-R Treatment

SUMMARY:
The proposed study will employ a cross-cultural Community Based Participatory Research (CBPR) approach to build from prior needs assessments and mixed-methods research to evaluate the effectiveness of the Family Strengthening Intervention for Refugees (FSI-R), a preventative family home-based visiting intervention intended to mitigate mental health disparities among refugee children and families using a hybrid implementation-effectiveness design. Results of the investigator's trial will expand the evidence-base on community-based interventions for refugees and has the potential to be replicated to reduce mental health disparities affecting diverse groups of refugee children and families.

DETAILED DESCRIPTION:
Using a CBPR approach, a family based prevention model, the Family Strengthening Intervention for Refugees (FSI-R) was adapted from a tested model used in Africa and designed for delivery by refugee community health workers with through a process involving stakeholder consultation and local refugee Community Advisory Board input. Pilot data on the FSI-R demonstrates strong feasibility and acceptability, but further data are needed on effectiveness as well as barriers and facilitators to implementation by community health workers embedded in refugee-serving social services agencies. Specific aims are to (1) examine the impact of a family-based preventive intervention on outcomes of parent-child relationships, family functioning, and child mental health using a Hybrid Type 2 Effectiveness-Implementation Design (families with children aged 7-17 in a two-arm randomized controlled trial); (2) identify barriers and facilitators to implementation of the FSI-R by community health workers by conducting a process evaluation concurrent with the delivery of the intervention; and (3) strengthen the science of community engagement to address health disparities by fortifying CBPR-based pathways of change via collaborative partnerships between refugee communities, service providers, and academic stakeholders.

ELIGIBILITY:
Inclusion Criteria for families:

* being a resettled refugee family
* having one or more school-aged children living in the home (aged 7-17)

Inclusion Criteria for parents/caregivers:

* be aged 18 or older
* cares for and lives in the same household of the children at least 50% of the time
* is the child'd legal guardian

Exclusion Criteria:

* not meeting the above inclusion criteria
* families in the midst of a crisis (e.g. active suicide attempts)

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in conflict via the Family Conflict Scale | T1 (Baseline), T2 (approximately 24-months post-baseline), T3 (6-months follow-up from T2)
  The Family Conflict Scale utilizes a 7-point Likert Scale (0-6) to assess family conflict within the past month. Higher scores reflect greater family conflict.
Change in communication via the Revised Parent- Adolescent Communication Form | T1 (Baseline), T2 (approximately 24-months post-baseline), T3 (6-months follow-up from T2)
  Utilizes a 5-point Likert scale (1-5) to assess parent-child communication. Greater scores indicate higher communication between parents and their children.
Change in family conflict via the Intergenerational Conflict Index | T1 (Baseline), T2 (approximately 24-months post-baseline), T3 (6-months follow-up from T2)
  Utilizes a 5-point Likert scale (1-5) to assess intergenerational congruence across several domains of the parent-child relationship. Higher scores denote greater intergenerational congruence.
Change in parenting via the Alabama Parenting Questionnaire | T1 (Baseline), T2 (approximately 24-months post-baseline), T3 (6-months follow-up from T2)
  Likert scale (1-5) that includes 5 sub-domains. Each sub-domain results in a summed score that relates to 5 domains of parenting: involvement, positive parenting, poor monitoring/supervision, inconsistent discipline, and corporal punishment.

SECONDARY OUTCOMES:
Change in youth externalizing behaviors via the African Youth Psychosocial Assessment | T1 (Baseline), T2 (approximately 24-months post-baseline), T3 (6-months follow-up from T2)
  This assessment utilizes a 4-point Likert scale (1-4) to assess for externalizing problems in youth with greater scores reflecting greater conduct problems.
Change in youth depression via the Center for Epidemiologic Studies-Depression scale | T1 (Baseline), T2 (approximately 24-months post-baseline), T3 (6-months follow-up from T2)
  This measures utilizes a 4-point Likert scale (0-3) to assess depression in youth with higher scores indicated increasing levels of depression. The time frame referenced is "during the past week".

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Betancourt, ScD, Principal Investigator — Boston College
Locations (2):
- United States (2):
  - Maine Immigrant and Refugee Services, Lewiston, Maine
  - Jewish Family Service, Springfield, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jung E, Black C, Placencio-Castro M, Chamlagai L, Osman R, Hoffman M, Beardslee W, Betancourt TS. Delivering a family-based child mental health promotion program among two resettled refugee communities during the COVID-19 pandemic: Lessons learned in a hybrid type II implementation-effectiveness randomized controlled trial. Am J Community Psychol. 2025 Oct 5. doi: 10.1002/ajcp.70021. Online ahead of print. PMID 41046558